CLINICAL TRIAL: NCT02281383
Title: Phase II Study to Evaluate the Response to 2 Induction Courses (12 Intravesical Instillations) of Bacillus Calmette-Guérin (BCG) for High Risk Superficial Bladder Cancer
Brief Title: Evaluate the Response to 2 Induction Courses (12 Intravesical Instillations) of Bacillus Calmette-Guérin (BCG) for High Risk Superficial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-174
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-02

CONDITIONS: Bladder Cancer; High Risk Superficial
Keywords: Bacillus Calmette-Guérin (BCG); 14-174
MeSH Terms: conditions — Urinary Bladder Neoplasms

ARMS (1):
- Bacillus Calmette-Guérin (BCG) (Experimental): Patients will be treated with an induction course (6 intravesical instillations) of BCG followed by a second induction course (6 intravesical instillations), with a recovery period between the 2 treatment courses.
  Interventions: Biological: Bacillus Calmette-Guérin (BCG)

INTERVENTIONS:
Biological: Bacillus Calmette-Guérin (BCG)

SUMMARY:
This is a phase II study. This means that BCG therapy has already been found to be safe in humans. The investigators just want to see if using more treatments works better.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have high risk non-muscle invasive urothelial bladder carcinoma (Tis, TaHG, or T1) that is pathologically confirmed by the Memorial Sloan Kettering Department of Pathology or a documented history of TaHG or T1 non-muscle invasive urothelial bladder tumors.
* 18 years and older
* All visible papillary lesions must be macroscopically resected within 60 days of treatment initiation.
* Absence of urothelial carcinoma involving the upper urinary tract (documented by radiological imaging or biopsy) preferably within 12 months from the start of treatment. Should the imaging or biopsy be performed outside this window it will be up to the physicians discretion to re-scan/biopsy.
* Patients who have received a single dose of mitomycin C following staging TUR.

Exclusion Criteria:

* Currently being treated or scheduled to have radiation treatment for bladder cancer during the study.
* Treatment with intravesical BCG or chemotherapy for a patient's current <T2 tumor during the 12 months prior to the current diagnosis.
* Currently being treated or scheduled to have treatment with any systemic or intravesical chemotherapeutic agent during the study.
* Currently being treated with or having been treated in the last 12 months with any investigational drug for high risk superficial bladder cancer.
* Previous muscle-invasive (i.e., stage T2 or higher) transitional cell carcinoma of the bladder.
* Currently being treated for metastatic transitional cell carcinoma.
* Scheduled to have surgery for bladder cancer during the study.
* Presence of clinically significant infections or congenital or acquired immunodeficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry W. Herr, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacillus Calmette-Guérin (BCG): Patients will be treated with an induction course (6 intravesical instillations) of BCG followed by a second induction course (6 intravesical instillations), with a recovery period between the 2 treatment courses.
  Bacillus Calmette-Guérin (BCG)
Period: Overall Study
Arm/Group | Bacillus Calmette-Guérin (BCG)
Started | 80
Completed | 68
Not Completed | 12
Not completed — Progressive Disease | 1
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 2
Not completed — Death | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bacillus Calmette-Guérin (BCG)
Number analyzed (Participants) | 80
Age, Continuous [Median (Full Range); unit: years] | 71 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 70
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: (by cystoscopy and cytology) Participants who have a response are those who have no evidence of disease in their bladder by both urine cytology and cystoscopy. Participants whose disease remains at the same stage or is downstaged without complete resolution are considered nonresponders and will be documented as having recurred. Participants with worsening tumor, defined as the upstaging from non-muscle invasive to muscle invasive disease, or metastatic disease will be documented as disease progression.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bacillus Calmette-Guérin (BCG)
Number analyzed (Participants) | 80
Participants
  Complete Response | 62
  Stable Response | 18

2. Secondary Outcome: Percentage of Participants With Recurrence-free Survival After Complete Response
Description: Progression is defined as the upstaging, from non-muscle invasive to muscle invasive disease, or metastatic disease will be documented as disease progression.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bacillus Calmette-Guérin (BCG)
Number analyzed (Participants) | 62
percentage of participants | 85 [77 to 95]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Bacillus Calmette-Guérin (BCG)
All-Cause Mortality (participants affected / at risk) | 8/80
Serious Adverse Events (participants affected / at risk) | 4/80
Other Adverse Events (participants affected / at risk) | 12/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bacillus Calmette-Guérin (BCG) (N=80)
Hematuria (Renal and urinary disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bacillus Calmette-Guérin (BCG) (N=80)
Fatigue (General disorders) | 8
Cystitis noninfective (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT02281383/Prot_SAP_000.pdf